CLINICAL TRIAL: NCT05523986
Title: Vitamin D Treatment Effect for Atopic Dermatitis in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC1-111
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; human microbiome; vitamin D; vitamin D receptors and vitamin D binding protein
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment group (Experimental): Vitamin D (2000IU/day) for 6 months
  Interventions: Other: Vitamin D
- Placebo Comparator: Control group (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Vitamin D (2000IU/day) for 6 months
  Arms: Experimental: Treatment group
Other: Placebo — Placebo
  Arms: Placebo Comparator: Control group

SUMMARY:
A double-blind study to evaluate the role of human microbiome and vitamin D in the development of atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic relapsing inflammatory skin disease with intermittent flares, affecting approximately 15% to 20% worldwide. Atopic dermatitis is clinically distinguished by pruritus, eczematous plaques, and a defective epidermal barrier. The pathology of AD is not entirely understood. It involves a complex interplay of dysfunctions of immune response, genetic and environmental factors (such as exposure to allergens and microbes). The control of patients with AD may be difficult to be achieved in some patients; this suggests the presence of some other associated factors. The findings obtained in both clinical and observational studies revealed that the deficiency of vitamin D may be a factor to be considered in the pathophysiology of AD. Vitamin D supplementation with standard treatment yielded positive clinical outcomes in mild and moderate AD. However, the potential benefit of vitamin D and its clinical correlation in AD is still uncertain. Thus, there is a need for more detailed and prospective studies.

The investigators will enroll children with atopic dermatitis and age and gender matched healthy children in China Medical University Children's Hospital. Briefly, the investigators interviewed subjects using EASI SCORE (defined as moderate or severe patients) and collected their venous blood and microbiome samples of nasal, skin and anal swab. Then, AD subjects will be given vitamin D or placebo for 6 months in a randomized, double-blind way. The participants will be asked to return to the outpatient clinic every month to assess the severity of AD. After six months of follow-up, their blood, nasal cavity, skin and intestinal bacterial samples were taken. All microbial analysis, allergen detection, vitamin D concentration, VDR, and DBP genotype will be analyzed by the core laboratory and bioinformatics center of CMUH.

The investigators believe this study can answer the cause-effect relationships of microbiota and vitamin D in the development of AD, and design a microbiota-related preventive and treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

Experimental group: Patients were 1-18 years old with EASI score moderate to severe atopic dermatitis, and atopic dermatitis was defined as three or more of the following statements to be diagnosed as atopic dermatitis:

1. skin itching
2. typical skin symptoms (including eczematous dermatitis or lichenified dermatitis) and location (mostly on the extensor side of the face and body in infants and young children, and on the flexor side of joints in adults)
3. chronic persistent or recurrent dermatitis for more than 6 months.
4. Individuals or family members with atopic constitution such as allergic rhinitis, asthma, atopic dermatitis or urticaria.

Control group:healthy children under the age of 18 (eg, healthy siblings of sick children).

Exclusion Criteria:

1. Less than 1 year old or more than 18 years old.
2. Patients with mild EASI severity of atopic dermatitis.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Levels of vitamin D | Month 0
  Vitamin D will be measured in a blood sample by ELISA to determine baseline status.
Levels of vitamin D | Month 6
  Vitamin D will be measured in a blood sample to follow the change from baseline in vitamin D level at month 6.
Single nucleotide polymorphism of vitamin D receptor and vitamin D binding protein | Month 0
  Single nucleotide polymorphism (SNP) genotyping will be performed in a blood sample by using TaqMan SNP genotyping assays.
Microbiome Microbiome | Month 0
  Nasal, skin and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome Microbiome | Month 6
  Nasal, skin and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing,and to follow the change from baseline in microbiome at month 6.
Total IgE | Month 0
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to determine baseline status.
Total IgE | Month 6
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to follow the change from baseline in total IgE at month 6.
Allergen-specific IgE | Month 0
  Plasma allergen-specific IgE will be measured by BioIC ®.

SECONDARY OUTCOMES:
The Eczema Area and Severity Index (EASI) | Month 0 to Month 6
  EASI range is from 0 to 72, the minimum value is "0" and maximum value is "72", higher scores mean a worse outcome.
Patient Oriented Eczema Measure (POEM) | Month 0 to Month 6
  This survey is a total of 7 questions that assesses the quality of life of patient's with eczema to determine their disease severity. The 7 questions are scored out of 4 points. A higher total score indicates a higher severity of disease.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan